CLINICAL TRIAL: NCT00006352
Title: The SILVA Study: Survival in an International Phase III Prospective Randomized LD Small Cell Lung Cancer Vaccination Study With Adjuvant BEC2 and BCG
Brief Title: Monoclonal Antibody Therapy Plus BCG in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-08971B; EORTC-08971B
Record Dates: First submitted 2000-10-04; First posted 2003-07-28 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — BCG Vaccine

INTERVENTIONS:
Biological: BCG vaccine
Biological: monoclonal antibody BEC2

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. BCG may activate the immune system to kill tumor cells. Combining monoclonal antibody therapy with BCG may kill more tumor cells. It is not yet known if monoclonal antibody therapy plus BCG is an effective treatment for limited-stage small cell lung cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of monoclonal antibody therapy plus BCG in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the impact of vaccination with adjuvant BCG and monoclonal antibody BEC2 on the survival of patients with limited stage small cell lung cancer.
* Determine the progression free survival in these patients after receiving this treatment regimen.
* Determine the safety of this treatment regimen in these patients.
* Assess the quality of life in these patients treated with this regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, Karnofsky performance status (60-70% vs 80-100%), and response to first line combined modality treatment (complete remission vs partial remission). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive vaccination with BCG and monoclonal antibody BEC2 intradermally on day 1 of weeks 0, 2, 4, 6, and 10 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive no further therapy. Quality of life is assessed at baseline; at weeks 6, 12, and 24; and every 6 months thereafter until disease progression.

Patients are followed at 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 570 patients (285 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed limited stage small cell lung cancer (SCLC)

  * Completed first line combination treatment consisting of at least a 2 drug chemotherapy regimen (4 to 6 courses) and a chest radiotherapy regimen

    * Must have achieved clinical response (complete or partial) with no evidence of progression or relapse

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* AST less than 1.5 times upper limit of normal
* No hepatitis B

Renal:

* Not specified

Other:

* No history of tuberculosis
* Purified Protein Derivative negative to at least 5 IU
* HIV negative
* No severe active infection
* No active infections requiring systemic antibiotics, antiviral, or antifungal treatments
* No serious unstable chronic illness
* No other prior malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or nonmelanomatous skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No prior therapy with mouse proteins
* No other concurrent immunotherapy before first disease progression

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy before first disease progression

Endocrine therapy:

* No concurrent systemic or chronic corticosteroids

Radiotherapy:

* See Disease Characteristics
* No prior radiation to spleen
* No concurrent radiotherapy before first disease progression

Surgery:

* No prior surgery for SCLC
* No prior splenectomy

Other:

* At least 4 weeks since prior combination therapy
* No prior second line therapy for SCLC
* At least 4 weeks since other prior investigational agent
* No concurrent systemic antihistamines or nonsteroidal antiinflammatory drugs
* No concurrent immunosuppressant therapy before first disease progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 1999-09; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center
Locations (1):
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands

REFERENCES:
- [Result] Giaccone G, Debruyne C, Felip E, Chapman PB, Grant SC, Millward M, Thiberville L, D'addario G, Coens C, Rome LS, Zatloukal P, Masso O, Legrand C. Phase III study of adjuvant vaccination with Bec2/bacille Calmette-Guerin in responding patients with limited-disease small-cell lung cancer (European Organisation for Research and Treatment of Cancer 08971-08971B; Silva Study). J Clin Oncol. 2005 Oct 1;23(28):6854-64. doi: 10.1200/JCO.2005.17.186. PMID 16192577